CLINICAL TRIAL: NCT05128955
Title: Embolization of the Splenic Artery After Trauma (ELSA-2)
Brief Title: Embolization of the Splenic Artery After Trauma
Acronym: ELSA-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew J. Gunn (Other)
Collaborators: Penumbra Inc. (Industry)
Responsible Party: Sponsor-Investigator, Andrew J. Gunn, Associate Professor, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300008343; 000533374 (Other Grant/Funding Number: Penumbra, Inc.)
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: High-grade Splenic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Comparator: Splenic artery embolization with vascular embolic coils (Active Comparator): Device: Splenic artery embolization with vascular embolic coils
  Interventions: Device: Splenic artery embolization with vascular embolic coils or plugs
- Active Comparator: Splenic artery embolization with vascular embolic plugs (Active Comparator): Active Comparator: Splenic artery embolization with vascular embolic plugs
  Interventions: Device: Splenic artery embolization with vascular embolic coils or plugs

INTERVENTIONS:
Device: Splenic artery embolization with vascular embolic coils or plugs — Splenic artery embolization with vascular embolic coils or plugs

SUMMARY:
Our aim is to conduct a multi-center, Bayesian, randomized clinical trial to evaluate the primary technical success of coils and vascular plugs for proximal splenic artery embolization in the setting of high-grade splenic trauma. The investigator has previously demonstrated the feasibility of such a study in a single center pilot trial.

DETAILED DESCRIPTION:
Splenic preservation rates are improved for participants with high-grade splenic injuries (defined as Grade III-V injuries by the American Association for the Surgery of Trauma (AAST) guidelines) when non-operative management is supplemented by image-guided, trans-catheter splenic artery embolization (SAE). SAE is currently the standard of care for hemodynamically stable participants with high-grade splenic injuries. In proximal SAE (pSAE), the mid-splenic artery is embolized between the origins of the dorsal pancreatic artery and pancreatica magna artery with either endovascular plugs (VPs) or endovascular coils (EC). This reduces the intra-splenic arterial pressure which allows the parenchyma time to heal. Splenic perfusion is maintained via a collateral pathway consisting of flow from the splenic artery proximal to the site of embolization through the smaller dorsal pancreatic artery to the transverse pancreatic artery to the pancreatica magna artery which then delivers a slower, smaller amount of blood to the splenic artery distal to the site of embolization. Additionally, collateral supply from the short gastric and gastroepiploic arteries helps to protect the spleen from infarction and/or abscess formation.

pSAE is most often accomplished using either VPs or ECs as the embolic agent, both of which are FDA-approved and clinically-available. ECs have a long history of efficacy and safety for embolization and are thus familiar embolic agents to most endovascular specialists. Further, coils large enough to embolize the mid-splenic artery can be deployed through a standard micro-catheter, which means they can be used in even the most tortuous splenic arteries. However, multiple coils may need to be deployed in the same patient to achieve hemostasis in the mid-splenic artery that may increase their overall cost, iodinated contrast use, procedural time, and the radiation exposure to the participant and medical staff. Additionally, given the high-flow nature of the splenic artery, even an appropriately sized coil may migrate distally. A typical pSAE using coils will involve the deployment of one helical coil followed by multiple packing coils until hemostasis is achieved. VPs attempt to overcome the limitations of coils. For example, the deployment of a single VP can typically provide hemostasis in the mid-splenic artery which theoretically reduces procedural time, contrast load, and radiation exposure. Despite this, VPs are usually more expensive than coils on a per unit basis and are usually less familiar devices to endovascular specialists. Another drawback of VPs is that they cannot be deployed through a standard micro-catheter but rather require the advancement of a larger, stiffer 0.035 inch system into the mid-splenic artery. This may limit their use in very tortuous splenic arteries. Currently, the selection of embolic agent for pSAE is primarily based on operator experience and preference. The embolic efficacy, technical success, and cost of using coils compared to VPs has been evaluated in other diseases; yet, to the best of our knowledge, these embolic agents have never been compared for their use in pSAE, much less in a randomized, prospective fashion.

ELIGIBILITY:
Inclusion Criteria:

1. ≥15 years of age
2. Trauma resulting in grade III or higher splenic injury on contrast-enhanced CT
3. Splenic injury to be treated by non-operative management as decided by attending trauma surgeon and interventional radiologist
4. The attending interventional radiologist determines that the patient will undergo proximal splenic artery embolization with the specific method to be decided by randomization.

Exclusion Criteria:

1. Inability to obtain informed consent
2. ≤ 50kg
3. Uncorrectable coagulopathy
4. Patient is immunocompromised
5. Pregnant
6. Breast-feeding
7. Non-English speakers
8. Prisoners

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary Technical Success | 3 years
  The ability to deploy the assigned embolic device in the mid-splenic artery with resultant occlusion of the artery within 15 minutes of deployment.

SECONDARY OUTCOMES:
Number of Participants Enrolled within 24 months | 24 months
  The primary outcome of the study will be to enroll 250 participants within 24 months of study initiation with adequate 30 day follow-up on all participants.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Prisma Health, Greenville, South Carolina
  - The University of Texas Health Science Center at Houston McGovern Medical School, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided